CLINICAL TRIAL: NCT01421641
Title: The Effect of Intracervical Lidocaine Injection Versus Topical Lidocaine Gel on the Pain Experienced by Patients Undergoing Tenaculum Application to the Cervix at the Time of an Office Gynecologic Procedure
Brief Title: Tenaculum Pain Control Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Paula Bednarek, MD MPH, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: OHSU RES 7148
Record Dates: First submitted 2011-08-09; First posted 2011-08-23 (Estimated); Results first posted 2014-04-21 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-03

CONDITIONS: Cervical Pain; Pelvic Pain
Keywords: Tenaculum; Pain; Lidocaine
MeSH Terms: conditions — Neck Pain; Pelvic Pain; Pain | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intracervical Lidocaine Injection (Active Comparator): Injection of 2 cc of 1% lidocaine solution at the anterior lip of the cervix using a standard 22 gauge spinal needle.
  Interventions: Drug: Intracervical Lidocaine Injection
- Topical Lidocaine Gel (Active Comparator): Application of 1cc of 2% lidocaine gel to the anterior lip of the cervix with a Q-tip (this amount of lidocaine will be measured out prior to procedure)
  Interventions: Drug: Topical Lidocaine Gel

INTERVENTIONS:
Drug: Intracervical Lidocaine Injection — Injection of 2 cc of 1% lidocaine solution at the anterior lip of the cervix using a standard 22 gauge spinal needle
  Other Names: Lidocaine injection, paracervical blocker
  Arms: Intracervical Lidocaine Injection
Drug: Topical Lidocaine Gel — Application of 1cc of 2% lidocaine gel to the anterior lip of the cervix with a Q-tip
  Other Names: lidocaine gel, numbing gel
  Arms: Topical Lidocaine Gel

SUMMARY:
The purpose of this clinical trial is to evaluate the effect of an intracervical lidocaine injection versus topical lidocaine gel on the pain experienced by patients undergoing tenaculum application to the cervix during office gynecologic procedures. This study will also evaluate how satisfied women are with the method of pain control used.

The researchers hypothesize that:

1. There is less pain perceived by patients undergoing placement of a tenaculum on the cervix when a lidocaine injection is used compared to a topical lidocaine gel.
2. Patients are more satisfied with pain control during the overall experience of undergoing tenaculum placement on the cervix when a lidocaine injection is used compared to a topical lidocaine gel.

DETAILED DESCRIPTION:
Subjects who have already scheduled an IUD insertion or endometrial biopsy will be asked to join this study assessing two pain control interventions at the time of tenaculum application to the cervix during office gynecologic procedures. Only healthy women ages 18 and over with an indication for endometrial biopsy or IUD placement will be recruited. The participants will be randomized to one of two arms: an intracervical lidocaine injection versus topical lidocaine gel. They will be asked to indicate their level of pain and level of satisfaction using a Visual Analog Scale. The primary outcome, pain with tenaculum placement, and the secondary outcome, satisfaction with the experience of tenaculum placement, will be compared between the study groups.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy women
* Age 18 and over
* Indication for endometrial biopsy or IUD placement

Exclusion Criteria:

* Allergy to lidocaine or other local anesthetic
* Pregnancy, known or suspected
* Patients who are premedicated with misoprostol
* Patients with a chronic pain condition for which the patient takes daily pain medication

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2011-09; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paula Bednarek, MD MPH, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We conducted a randomized, single-blinded clinical trial from August 2011 to May 2012 at the Center for Women's Health at Oregon Health & Science University (OHSU; Portland, Oregon).We recruited women aged 18 years and older who were scheduled to undergo IUD placement or endometrial biopsy.
Pre-assignment Details: Exclusion criteria included 1) allergy to lidocaine or other local anesthetics; 2) pregnancy; 3) patients pre-medicated with misoprostol; and 4) patients with a chronic pain condition for which they were taking daily pain medications of any kind. The subjects were recruited, consented, and enrolled immediately prior to the procedure.
Groups:
- Intracervical Lidocaine Injection: Intracervical Lidocaine Injection : Injection of 2 cc of 1% lidocaine solution at the anterior lip of the cervix using a standard 22 gauge spinal needle
- Topical Lidocaine Gel: Topical Lidocaine Gel : Application of 1cc of 2% lidocaine gel to the anterior lip of the cervix with a Q-tip
Period: Overall Study
Arm/Group | Intracervical Lidocaine Injection | Topical Lidocaine Gel
Started | 37 | 37
Completed | 35 | 35
Not Completed | 2 | 2
Not completed — Protocol Violation | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intracervical Lidocaine Injection | Topical Lidocaine Gel | Total
Number analyzed (Participants) | 37 | 37 | 74
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 37 | 37 | 74
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.6 (12.2) | 33.7 (7.3) | 34.5 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 37 | 74
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 37 | 37 | 74

OUTCOME MEASURES:

1. Primary Outcome: Tenaculum Pain
Description: The primary outcome was pain at the time of tenaculum placement. Patient asked to pain scale using 100mm Visual Analog Scale (0mm=no pain, 100mm=worst pain of my life) during after tenaculum placement.
Time Frame: After tenaculum placement
Population: 4 subjects were excluded due to protocol violations
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Intracervical Lidocaine Injection | Topical Lidocaine Gel
Number analyzed (Participants) | 35 | 35
mm | 12.3 (17.4) | 36.6 (23.0)

2. Secondary Outcome: Intervention Pain
Description: Pain with the intervention (injection or gel application). Subjects are asked to complete pain scale using a 100mm Visual Analog Scale (0mm=no pain and 100mm=worst pain of my life)
Time Frame: after application of randomized intervention
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Intracervical Lidocaine Injection | Topical Lidocaine Gel
Number analyzed (Participants) | 35 | 35
mm | 20.4 (19.4) | 5.9 (8.6)

3. Secondary Outcome: Tenaculum Placement Satisfaction
Description: Satisfaction with overall tenaculum placement procedure. Subjects asked to answer their overall satisfaction with the pain control. Subjects asked to complete 100mm Visual Analog Scale (0mm=not at all satisfied to 100mm=very satisfied)
Time Frame: After placement of the tenaculum
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Intracervical Lidocaine Injection | Topical Lidocaine Gel
Number analyzed (Participants) | 35 | 35
mm | 79.9 (22.7) | 74.6 (27.6)

ADVERSE EVENTS:
Arm/Group | Intracervical Lidocaine Injection | Topical Lidocaine Gel
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/37
Other Adverse Events (participants affected / at risk) | 1/37 | 0/37
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Intracervical Lidocaine Injection (N=37) | Topical Lidocaine Gel (N=37)
vasovagal reaction (Nervous system disorders) | 1 (1) | 0/36 (0) — After completion of the tenaculum study portion of the procedure, the patient had a vasovagal reaction at the time of insertion of the intrauterine device. This is not likely to be related to the study intervention, and resolved completely.

LIMITATIONS AND CAVEATS:
There are several limitations to this study, including potential selection bias, difficulty with blinding the intervention, timing of the intervention for maximal effect, and the limitations inherent in measuring pain.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No